CLINICAL TRIAL: NCT02108418
Title: A Phase 1, Randomized, Open-label, 2-way Crossover Study in Healthy East Asian and Caucasian Volunteers to Evaluate the Relative Bioavailability of A New Capsule Formulation of TG-2349 Compared to the Original Formulation of TG-2349 Oral Solution
Brief Title: Study to Evaluate the PK, Relative Bioavailability and Safety of TG-2349 With Single Oral Dose Under Fed Condition in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TaiGen Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: TG-2349-02
Record Dates: First submitted 2014-03-27; First posted 2014-04-09 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Healthy
MeSH Terms: interventions — Dosage Forms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TG-2349 as the original formulation (Experimental): 400 mg, 2 syringes
  Interventions: Drug: TG-2349 as the original formulation
- TG-2349 as a new capsule formulation (Experimental): 400 mg, 4 capsules
  Interventions: Drug: TG-2349 as a new capsule formulation

INTERVENTIONS:
Drug: TG-2349 as the original formulation — single oral dose under fed condition
  Arms: TG-2349 as the original formulation
Drug: TG-2349 as a new capsule formulation — single oral dose under fed condition
  Arms: TG-2349 as a new capsule formulation

SUMMARY:
1. To evaluate the pharmacokinetics (PK) and relative bioavailability of TG-2349, given as a new capsule formulation and as the original formulation of oral solution, after a single oral dose of 400 mg under fed condition in healthy volunteers.
2. To evaluate the safety and tolerability of TG-2349 in healthy volunteers.
3. To evaluate the ethnic differences in PK and safety between East Asian and Caucasian volunteers.

DETAILED DESCRIPTION:
TG-2349 oral solution has been investigated in a phase I/IIa study (study number: TG-2349-01) in healthy volunteers and patients with chronic hepatitis C (CHC) infection. The study demonstrated that TG-2349 was safe and well-tolerated when given to healthy volunteers at single oral doses up to 800 mg, and at five-consecutive daily oral doses up to 600 mg. Co-administration of TG-2349 with food resulted in a significant increase in bioavailability, and therefore concomitant food intake with dosing is recommended.

To further advance the clinical development of TG-2349, a new capsule formulation was developed to replace the current TG-2349 oral solution. The objectives of this study (study number: TG-2349-02) are to evaluate the PK and relative bioavailability of TG-2349, given as a new capsule formulation and as the original formulation of oral solution, after a single oral dose of 400 mg under fed condition in healthy volunteers, and to evaluate the safety, tolerability, and ethnic differences of the TG-2349 capsule formulation.

ELIGIBILITY:
Inclusion Criteria at Screening

1. East Asian or Caucasian subjects, male or female, and 18 to 40 years of age inclusive
2. Body mass index (BMI) in the range of 19.0 to 30.0 kg/m2 and body weight ≥ 50 kg inclusive
3. In general good physical and mental health status on the basis of a medical history review, medical evaluation including vital signs and physical examination, 12-lead ECG, and laboratory results at screening
4. For females, one of the following criteria must be fulfilled:

(1)At least 1 year post menopausal, or (2)Surgically sterile, or (3)Willing to use a double-barrier method (intrauterine device [IUD] plus condom, spermicidal gel plus condom) of contraception from screening until 30 days after the last dose of study drug; 5.Males must be willing to use a reliable form of contraception (use of a condom or a partner fulfilling the above criteria) from screening until 30 days after the last dose of study drug 6.Willing to abstain from caffeine- or xanthine-containing beverages (including coffee and tea), alcohol, grapefruit juice, and Seville oranges during the stay-on-site period 7.Willing and able to provide written informed consent

Exclusion Criteria at Screening

1. Positive serological test for IgM anti-HAV antibody, HbsAg, or anti-HCV antibody at screening
2. Positive ELISA test for HIV-1 or HIV-2 at screening
3. Any of the following abnormal laboratory values at screening: Hemoglobin (Hb) <12.0g/dL for women and <13.0g/dL for men, white blood cell count (WBC) <3,000 cells/mm3, absolute neutrophil count <1,500 cells/mm3, platelet count <100,000 cells/mm3, serum creatinine ≥ 2 mg/dL, ALT or AST levels ≥ 2 xULN, total bilirubin ≥ 1.5 xULN, INR (International Normalized Ratios for prothrombin time) ≥1.5 xULN
4. Any abnormal laboratory values that are considered clinically significant by the Investigator at screening
5. QTcF greater than 450 msec for females and 430 msec for males at screening
6. History of renal, hepatic impairment, stomach or intestinal surgery or resection, malabsorption syndrome
7. History of seizures, epilepsy, cardiovascular, diabetes, or cancer (except basal cell carcinoma)
8. History or family history of prolonged QT interval or family history of sudden cardiac death at a young age (< 30 years )
9. History of drug allergy or hypersensitivity, especially to sulfa drugs
10. History or evidence of abuse of alcohol, barbiturate, amphetamine, recreational, or narcotic drug use within 6 months prior to first dose of study drug administration
11. Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of a psychiatric illness, or who have any history of suicide attempt or depression
12. Anemia or blood/plasma donation within 30 days prior to first dose of study drug administration
13. Pregnant or breast-feeding
14. Use of tobacco or nicotine-containing products within 30 days prior to first dose of study drug administration
15. Use of concomitant medication, including herbal remedies and dietary supplements (except for paracetamol/acetaminophen, ibuprofen, and hormonal contraceptives) within 14 days prior to first dose of study drug administration
16. Received any other investigational drug within 30 days prior to first dose of study drug administration

Exclusion Criteria at the First Admission

1. Any of the following abnormal laboratory values at admission: Hb <12.0g/dL for women and <13.0g/dL for men, WBC <3,000 cells/mm3, absolute neutrophil count <1,500 cells/mm3, platelet count <100,000 cells/mm3, serum creatinine ≥ 2 mg/dL, ALT or AST levels ≥ 2 xULN, total bilirubin ≥ 1.5 xULN, INR ≥ 1.5 xULN
2. Any abnormal laboratory values that are considered clinically significant by the Investigator at admission
3. Any clinically significant abnormality on 12-lead ECG or a QTcF greater than 450 msec for females and 430 msec for males at admission
4. Positive urine drug screen or breath alcohol test at admission
5. If female, positive serum pregnancy test at admission
6. Acute illness within 2 weeks prior to dosing, unless approved by the Sponsor's Medical Monitor

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-04; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Primary pharmacokinetic parameters: AUC0-t, AUC0-inf and Cmax | 120 hours after administration of study drug in each session

SECONDARY OUTCOMES:
Secondary pharmacokinetic parameters:Tmax, t1/2, CL/F, V/F and λz | 120 hours after administration of study drug in each session
Urine pharmacokinetic parameters: Urine Ae% | 120 hours after administration of study drug in each session
Stool pharmacokinetic parameters: Stool Ae% | 120 hours after administration of study drug in each session
Safety parameters: Incidence and severity of AEs, changes from baseline in safety laboratory values, 12-lead ECG parameters, vital signs, and physical examination. | approximately 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Sims, DO, Principal Investigator — WCCT
Locations (1):
- WCCT, Cypress, California, United States